CLINICAL TRIAL: NCT06017284
Title: Thalidomide to Chemotherapy Related Nausea and Vomiting in Pancreatic Cancer
Acronym: PTCA199-5
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Guopei Luo, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PTCA199-5
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Pancreatic Cancer Stage IV; Chemotherapy-induced Nausea and Vomiting
Keywords: chemotherapy; pancreatic cancer; Thalidomide; nausea; quality of life
MeSH Terms: conditions — Pancreatic Neoplasms; Vomiting; Nausea | interventions — Thalidomide; Taxes; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemotherapy + Thalidomide (Experimental): nab-paclitaxel (120 mg per square meter of body-surface area) followed by gemcitabine (1000 mg per square meter) on days 1, 8, and 15 every 4 weeks. Thalidomide 100 mg/day, once a day, orally intake at night.
  Interventions: Drug: Thalidomide; Drug: Nab paclitaxel; Drug: Gemcitabine
- Chemotherapy (Active Comparator): nab-paclitaxel (120 mg per square meter of body-surface area) followed by gemcitabine (1000 mg per square meter) on days 1, 8, and 15 every 4 weeks.
  placebo 100 mg/day, once a day, orally intake at night.
  Interventions: Drug: Nab paclitaxel; Drug: Gemcitabine; Drug: Placebo

INTERVENTIONS:
Drug: Thalidomide — Thalidomide 100 mg/day, once a day, orally intake at night.
  Arms: Chemotherapy + Thalidomide
Drug: Nab paclitaxel — nab-paclitaxel (120 mg per square meter of body-surface area) on days 1, 8, and 15 every 4 weeks.
Drug: Gemcitabine — gemcitabine (1000 mg per square meter) on days 1, 8, and 15 every 4 weeks.
Drug: Placebo — Placebo, 100 mg/day, once a day, orally intake at night.
  Arms: Chemotherapy

SUMMARY:
The purpose of this study is to evaluate the efficacy of thalidomide on improving the quality of life for metastatic pancreatic cancer patients receiving gemcitabine and nab-paclitaxel chemotherapy.

DETAILED DESCRIPTION:
Pancreatic cancer is a highly lethal malignancy with a 5-year survival less than 10%. Approximately 80% of patients with pancreatic cancer are diagnosed at an advanced stage. Chemotherapy is one of the major treatments for advanced pancreatic cancer. The Metastatic Pancreatic Cancer Trial (MPACT) has confirmed the efficacy of gemcitabine combined with nab-paclitaxel as the first-line treatment to metastatic pancreatic cancer. However, the side-effects related to gemcitabine combined with nab-paclitaxel including nausea/vomiting, insomnia, fatigue, nausea, and malnutrition have impaired the tolerability of the regimen.

Thalidomide is an oral medication used to treat a number of cancers (e.g. multiple myeloma), graft-versus-host disease, and many skin disorders (e.g. complications of leprosy such as skin lesions). It caused severe malformations in babies born to mothers taking the drug for morning sickness in the late 1950s and early 1960s. Thalidomide works on the immune system to reduce inflammation. Thalidomide may enhance the tolerability of chemotherapy by reducing nausea/vomiting, improving sleeping quality, alleviating pain, and thus improving quality of life for patients with pancreatic cancer.

The purpose of this study is to evaluate the efficacy of Thalidomide on improving the quality of life for metastatic pancreatic cancer patients receiving gemcitabine and nab-paclitaxel chemotherapy. One hundred patients will be randomly assigned to the experimental group (gemcitabine combined with nab-paclitaxel, Thalidomide) or the control group (gemcitabine combined with nab-paclitaxel). Rate of nausea/vomiting, index of sleep quality, severity of pain, quality of life, and overall survival are measured every four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document.
* Age ≥ 18 years and ≤ 80 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Histologically or cytologically confirmed metastatic pancreas adenocarcinoma.
* Adequate organ performance based on laboratory blood tests.
* Presence of at least of one measurable lesion in agreement to Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* The expected survival ≥ 3 months.
* Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation.

Exclusion Criteria:

* Patients who have received any form of anti-tumor therapy.
* The diagnosis was confirmed by pathology as non-adenocarcinoma of pancreas.
* Inflammation of the digestive tract, including pancreatitis, cholecystitis, cholangitis, etc.
* Pregnant or nursing women.
* Severe and uncontrollable accompanying diseases that may affect protocol compliance or interfere with the interpretation of results, including active opportunistic infections or advanced (severe) infections, and diabetes that cannot be controlled after adequate clinical anti-hyperglycemia treatment according to guidelines, uncontrollable hypertension, cardiovascular disease (Class III or IV heart failure as defined by the New York Heart Association classification, congestive heart failure (CHF), myocardial infarction in the past 6 months , unstable arrhythmia or unstable angina, cerebral infarction within 3 months, etc).
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to gemcitabine, nab-paclitaxel, or other agents used in the study.
* Other serious accompanying illnesses, which, in the researcher's opinion, could seriously adversely affect the safety of the treatment.
* Patients who are unwilling or unable to comply with study procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Rate of nausea/vomiting | At the end of Cycle 1 (each cycle is 28 days)
  Rate of nausea/vomiting after every cycle of chemotherapy using the 4-point Likert scale. The range of scale is 0-3 and higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Pain numeric rating scale (NRS) | At the end of Cycle 1 (each cycle is 28 days)
  Change of pain numeric rating scale after every cycle of chemotherapy. The administration of analgesic drugs after every cycle of chemotherapy is recorded. The range of NRS scale is 0-10 and higher scores mean a worse outcome.
Quality of life (QOL) | At the end of Cycle 1 (each cycle is 28 days)
  Change of QOL after every cycle of chemotherapy assessed using European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30)
Sleep quality index | At the end of Cycle 1 (each cycle is 28 days)
  Sleep quality index after every cycle of chemotherapy is assessed using Pittsburgh sleep quality index (PSQI)
Overall survival (OS) | At the end of Cycle 1 (each cycle is 28 days)
  OS of subjects from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Guopei Luo, MD, Principal Investigator — Fudan University
Locations (1):
- Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang L, Qu X, Teng Y, Shi J, Yu P, Sun T, Wang J, Zhu Z, Zhang X, Zhao M, Liu J, Jin B, Luo Y, Teng Z, Dong Y, Wen F, An Y, Yuan C, Chen T, Zhou L, Chen Y, Zhang J, Wang Z, Qu J, Jin F, Zhang J, Jin X, Xie X, Wang J, Man L, Fu L, Liu Y. Efficacy of Thalidomide in Preventing Delayed Nausea and Vomiting Induced by Highly Emetogenic Chemotherapy: A Randomized, Multicenter, Double-Blind, Placebo-Controlled Phase III Trial (CLOG1302 study). J Clin Oncol. 2017 Nov 1;35(31):3558-3565. doi: 10.1200/JCO.2017.72.2538. Epub 2017 Aug 30. PMID 28854065
- [Background] Hwu WJ, Krown SE, Menell JH, Panageas KS, Merrell J, Lamb LA, Williams LJ, Quinn CJ, Foster T, Chapman PB, Livingston PO, Wolchok JD, Houghton AN. Phase II study of temozolomide plus thalidomide for the treatment of metastatic melanoma. J Clin Oncol. 2003 Sep 1;21(17):3351-6. doi: 10.1200/JCO.2003.02.061. PMID 12947072